CLINICAL TRIAL: NCT06999967
Title: Stanford-Lucidify Delirium Monitoring Pilot Study
Brief Title: Stanford-Lucidify EEG Delirium Study
Status: Not yet recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jose R Maldonado, MD, Medical Psychiatry Laboratory Director, Stanford University
Other Study IDs: 81015
Record Dates: First submitted 2025-05-16; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Delirium; Cognitive Dysfunction
Keywords: Delirium; EEG; Encephalopathy; Cognitive Dysfunction; Electroencephalography; Delirium Monitoring
MeSH Terms: conditions — Delirium; Cognitive Dysfunction; Brain Diseases | interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICU Population: Subjects admitted to the Intensive Care Unit (ICU)
  Interventions: Diagnostic Test: Electroencephalogram (EEG)
- Oncology Population: Subjects admitted to oncology units with hematologic malignancies undergoing cellular therapies or hematopoietic stem cell transplants (e.g., stem cell and Chimeric Antigen Receptor T-cell (CAR-T) Therapy)
  Interventions: Diagnostic Test: Electroencephalogram (EEG)

INTERVENTIONS:
Diagnostic Test: Electroencephalogram (EEG) — All study subjects will undergo monitoring via a portable electroencephalogram (pEEG), the CGX EEG system (a Research-grade 2-Channel EEG device) to measure the brainwaves of patients admitted to Stanford Medical Center. Investigators will then use the Lucidify software to allow for the interpretation of obtained brainwaves for the detection of delirium .

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the CGX/Lucidify EEG system in enabling physicians to detect delirium (confusion) in medically ill patients as early as possible in order to minimize the detrimental effects of delirium. The study will involve collecting EEG data through the CGX EEG system (a Research-grade 2-Channel EEG device) and applying the Lucidify EEG software algorithm to identify indicators and degree of delirium, obtain data regarding the amount and degree of patient's movement and activity throughout the day in order to detail delirium subtype, and obtain data regarding the quality of the sleep as it affects delirium severity and duration. By enhancing early detection, this research aims to improve patient outcomes and inform clinical decision-making.

DETAILED DESCRIPTION:
Study investigators would like to use a portable electroencephalogram (pEEG), the CGX EEG system (a Research-grade 2-Channel EEG device) to measure the brainwaves of patients admitted to Stanford Medical Center. Study investigators will then use the Lucidify software to allow for the interpretation of obtained brainwaves in order to detect delirium as early as possible, in order to minimize the detrimental effects of delirium in cognition and behavior. The Lucidify algorithm, different from our previously utilized EEG system (see below for details) can provide two additional features not previously available: (1) accelerometer data (an indicator of the level of patient's movements and a proxy for delirium phenotype; and (2) scored polysomnography data (providing validated interpretation of the patient's spectral sleep - thus a true measure of the patient's various stages and quality of sleep; which has direct implications on both the progression of delirium and the patient's overall health and recovery). Finally, the CGX system is simpler, more comfortable to wear, and better tolerated by medically ill patients.

The primary objective is to monitor the development and progression of delirium (acute confusion) and sleep disturbances associated with medical illness over time. The study will focus on two distinct patient populations: 1) patients admitted to an adult intensive care unit (ICU), and 2) patients in oncology units with hematologic malignancies undergoing cellular therapies or hematopoietic stem cell transplants (e.g., stem cell and Chimeric Antigen Receptor T-cell (CAR-T) Therapy). The rationale for targeting the occurrence of delirium, as its development has been associated with significantly poor hospital care outcomes and increased morbidity (medical complications) and mortality (death). The two patient populations have been specifically selected for the following reasons: Delirium is frequently observed in the ICU setting, with a reported prevalence of up to 85%. In the hematologic malignancies undergoing cellular therapies or hematopoietic stem cell transplants population, there is a significant prevalence of neurotoxicity associated with delirium, ranging from 20% to 60%. This neurotoxicity can lead to comorbid risks such as seizures and cerebral edema, and it is also associated with long-term cognitive impairment and depression (Hayden 2022, Ruark 2020).

In comparison to other portable EEG devices, the CGX EEG system investigators intend to investigate during the course of this specific study is more user-friendly (i.e., smaller, more portable, and has no wirings attaching the patient to the bed or an external device) , allowing for continuous monitoring without patient discomfort or interference associated with other monitoring systems currently used in our ICU setting. In addition to this system's tolerability and simplicity, this new device and AI-algorithm allows for the acquisition of two significant variables not previously available: (a) its algorithm allows for accelerometer data acquisition (this is a measure of the patient's motion, which will constitute an ideal and objective measure of the delirium phenotype (e.g., hypoactive, hyperactive, or mixed delirium subtype); and (b) the system allows for the measurement of the various phases of the sleep cycle, thus providing a full hypnogram of the quality and duration of sleep. Taking advantage of the enhanced comfort of wearing this new system; given the waxing and waning nature of delirium (i.e., how quickly it can vary through the course of 24-hrs) and In order to take full advantage of the system's capabilities, study investigators need the CGX recorder to remain in place 24/7 for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age is 55 years or older
2. Clinical suspicion of delirium or subject at risk for delirium
3. Admitted to the Intensive Care Unit (ICU) or Oncology wards
4. Expected hospital stay is greater than one (1) day
5. Subject must be fluent in English

Exclusion Criteria:

1. Age is younger than 55 years
2. Subjects with a primary neurological or neurosurgical condition such as stroke, epilepsy, brain tumor, or witnessed seizures, Parkinson's disease, traumatic brain injury, or s/p craniectomy
3. Active CNS substance abuse, intoxication, or withdrawal
4. Unarousable or unresponsive subjects with RASS <-3
5. Subject is blind, deaf, or unable to speak or understand English

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects admitted to the ICU or Oncology hospital wards
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with delirium accurately diagnosed by the CGX EEG/Lucidify System | 24-hours a day monitoring for a minimum of 3 days from enrollment to the end of the study period (maximum of 7 days post-enrollment)
  Record and collect EEG brain waves on study subjects using the CGX EEG/Lucidify System to assess EEG features to differentiate between delirium positive and delirium negative patients.
Development of Delirium | From enrollment to the end of the study period (maximum of 7 days post-enrollment)
  Number of subjects diagnosed with delirium
Determination of Delirium Phenotype | From enrollment to the end of the study period (maximum of 7 days post-enrollment)
  For those who develop delirium, the phenotype of delirium will be determined as per the Liptzin-Levkoff Criteria (based on DSM diagnostic Criteria). As such, all delirium episodes will be categorized as: hyperactive, hypoactive, mixed, or subsyndromal delirium. In addition, this phenotype determination will be compared with the CGX/Lucidify EEG System accelerometer data to determine concordance between the two.

SECONDARY OUTCOMES:
Immediate Post-hospital Admission Mortality | From date of admission up to time of discharge (assessed up to 1 year after admission)
  Mortality following admission to the ICU or oncology wards
Length of ICU & Hospital Stay | From date of admission up to time of discharge of the ICU or oncology ward, and then from the hospital (assessed up to 1 year after admission)
  Total number of days admitted to the hospital
Polysomnography Sleep Metrics - Stages of Sleep | 24 hours a day for a maximum of 7 days
  Assessment of the quality of the various sleep stages.
Polysomnography Sleep Metrics - Depth of sleep | 24 hours a day for a maximum of 7 days
  Assessment of the quality of the depth of sleep.
Polysomnography Sleep Metrics - Duration of Sleep | 24 hours a day for a maximum of 7 days
  Assessment of the duration of sleep.
Accelerometry Metrics - Acceleration Magnitude | 24 hours a day for a maximum of 7 days
  Assessment of the overall acceleration experienced by the device, useful for assessing movement intensity to measure the amount and degree of patient motion as a proxy for delirium motoric phenotype.
Accelerometry Metrics - Activity Counts | 24 hours a day for a maximum of 7 days
  Assessment of the number of subject movement events detected.
Accelerometry Metrics - Frequency of Movement | 24 hours a day for a maximum of 7 days
  Assessment of the rate at which movements occur, which can indicate activity patterns specific to a delirium motoric phenotype.
Accelerometry Metrics - Duration of Activity | 24 hours a day for a maximum of 7 days
  Assessment of the total time spent in different activity states, which can be indicative of a specific delirium motoric phenotype.
Accelerometry Metrics - Movement Variability | 24 hours a day for a maximum of 7 days
  Assessment of the variability in movement patterns, which can be indicative of a delirium motoric phenotype.

CONTACTS AND LOCATIONS:
Overall Officials: José R Maldonado, M.D., Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital and Clinics, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No